CLINICAL TRIAL: NCT04003285
Title: Novel Regenerative Therapeutic in Chronic Complex TBI
Brief Title: Allopregnanolone in Chronic Complex Traumatic Brain Injury
Acronym: ALLO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2798-I
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury (TBI)
Keywords: Brain Injuries, Traumatic; Depression; Pain
MeSH Terms: conditions — Brain Injuries, Traumatic; Depression; Pain | interventions — Pregnanolone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive 0 nM ALLO (placebo), 50 nM ALLO (lower dose ALLO) or 150 nM ALLO (higher dose ALLO).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, double-blind, placebo-controlled trial. All roles will be masked with the exception of the research pharmacist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Experimental): ALLO 0 nM (placebo: loading dose, 4-hour infusion, taper)
  Interventions: Drug: Placebo
- ALLO 50 nM (Experimental): ALLO 50 nM (lower dose ALLO: loading dose, 4 hour infusion, taper)
  Interventions: Drug: Allopregnanolone
- ALLO 150 nM (Experimental): ALLO 150 nM (higher dose ALLO: loading dose, 4 hour infusion, taper)
  Interventions: Drug: Allopregnanolone

INTERVENTIONS:
Drug: Placebo — ALLO 0 nM (placebo: loading dose, 4-hour infusion, taper)
  Arms: Placebo
Drug: Allopregnanolone — ALLO 50 nM (lower dose ALLO: loading dose, 4 hour infusion, taper)
  Arms: ALLO 50 nM
Drug: Allopregnanolone — ALLO 150 nM (higher dose ALLO: loading dose, 4 hour infusion, taper)
  Arms: ALLO 150 nM

SUMMARY:
This study will determine if allopregnanolone (ALLO) improves depression and pain symptoms in patients who have a history of mild traumatic brain injury (TBI) [primary endpoints]. The investigators will also determine if ALLO improves functional outcome [secondary endpoint]. Participants in this study will receive an intravenous infusion of either ALLO or placebo. Behavioral assessments will be conducted during the infusion and at several time points post-infusion.

DETAILED DESCRIPTION:
ALLO is a neurosteroid that exhibits multiple actions highly relevant to the treatment of chronic complex TBI. The investigators' recent human data suggest that ALLO is decreased in patients with TBI, suggesting that ameliorating deficits of this neurosteroid may be clinically therapeutic. In addition, multiple groups have reported ALLO reductions in patients with conditions that frequently co-occur with TBI, including depression and pain disorders. 132 Veterans with a history of mild TBI with co-occurring depression and pain symptoms (chronic complex TBI) will be randomized to either intravenous placebo or ALLO (3 groups/44 participants per group: placebo, lower dose ALLO, higher dose ALLO). Following a loading dose, Veterans will receive placebo or ALLO infusion targeted to achieve serum ALLO levels of 0 nM (placebo), 50 nM (ALLO lower dose), or 150nM (ALLO higher dose). Behavioral assessments will be conducted during the infusion, post-taper, and 24 hours post-infusion. In addition, the investigators will conduct behavioral assessments 7 days and 14 days post-infusion.

The investigators hypothesize that ALLO will be well-tolerated in patients with complex TBI, and that this intervention may reduce depression and pain symptoms (in addition to potentially improving function).

ELIGIBILITY:
Inclusion Criteria:

* 21-62 years of age, any ethnic group, either sex
* History of mild TBI since 2001 and service in the U.S. Military since 9/11/01 (OEF/OIF/OND era)
* The investigators will adhere to the operational definition of mild TBI suggested by the World Health Organization Task Force, with the exception of seizure and Glasgow Coma Scale score criteria (not available for these participants) with 1 or more of the following:

  * confusion or disorientation
  * loss of consciousness for 30 minutes or less
  * post-traumatic amnesia for less than 24 hours
  * and/or other transient neurological abnormalities such as focal signs, and intracranial lesion not requiring surgery
* Ability to participate fully in the informed consent process
* HAM-D score 14 (HAM-D range for moderate depression=14-18)
* Participants will meet DSM-5 criteria for major depressive disorder (by SCID)

  * The presence of psychotic features will be exclusionary
  * Single episodes or recurrent episodes will be permissible for study entry (the investigators will examine treatment responses in those who have had single depressive episodes versus those who have had multiple depressive episodes in exploratory sensitivity analyses
* BPI (Brief Pain Inventory, Short Form) 'current' pain intensity rating item score 4 (scale of 0-10)

  * Pain must be musculoskeletal in nature
* No anticipated need to alter psychiatric medications for 14-day duration of study involvement
* No changes in psychotropic or behavioral interventions during the study or in the 2 weeks prior to study enrollment
* Concomitant medications for co-occurring medical conditions are permissible for stable medical conditions that are reasonably well-controlled

  * for example, hypertension medications, statins, and oral hypoglycemic medications would generally be permissible if they appear to be effectively treating the underlying condition

Exclusion Criteria:

* Participants with current suicidal or homicidal ideation necessitating clinical intervention or representing an imminent concern
* Medications that could potentially confound study outcomes (for example, prednisone) are exclusionary
* Current DSM-5 diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition other than TBI
* Female participants who are pregnant or breast-feeding
* Known allergy to study medication
* Benzodiazepine, barbiturate, or opioid use within the last 2 weeks is exclusionary
* Substance use disorder (DSM-5), other than nicotine use disorder
* A serious medical illness, defined as an illness that requires hospitalization for additional care at the time of screening or one that has required hospitalization in the last month.

  * Any co-occurring medical illness should have a history of stable outpatient management
* Report of a history of seizures, a history of stroke, a history of prostate cancer (or any other cancer other than non-melanoma skin cancer), a history of myocardial infarction, the presence of congestive heart failure, or any other serious health condition that would likely preclude safe study participation in the medical opinion of the PI or in consultation with the participant's PCP/other health care provider
* Use of oral contraceptives, a hormone-releasing IUD, or other hormonal supplementation such as estrogen or progesterone, as there is a theoretical risk that a metabolite such as ALLO could potentially impact efficacy of oral contraceptives or estrogen replacement

Ages: 21 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory, Short Form (BPI-SF) Change | 6 hours, 24 hours, 7 days, and 14 days
  The Brief Pain Inventory, Short Form (BPI-SF) is a self-reported scale that measures the severity of pain and the interference of pain on function. The scores range from 0 (no pain) to 10 (pain as severe as you can imagine). There are 4 questions assessing worst pain, least pain, average pain in the past 24 hours, and pain right now. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
Hamilton-Depression Inventory (HAM-D) Change | 6 hours, 24 hours, 7 days, and 14 days
  The HAM-D measures the severity of depressive symptoms. It is a checklist of 17 items that are ranked on a scale of 0-4 or 0-2. The range for the total score (which is the sum of the scores of all 17 items) is 0-52; a higher score indicates greater severity of symptoms.

SECONDARY OUTCOMES:
Short Form Health Survey (SF-36) Change | 6 hours, 24 hours, 7 days, and 14 days
  The SF-36 is a health survey with an 8-scale profile embedded in 36 questions that measures physical and mental components of health. Each item is scored on a 0 to 100 range with the lowest and highest possible scores are set at 0 and 100, respectively. All of these items are scored so that a high score defines a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Christine E. Marx, MD MA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No